CLINICAL TRIAL: NCT00312273
Title: Aminophylline in Bradyasystolic Cardiac Arrest: A Randomized Placebo-Controlled Trial
Brief Title: Aminophylline in Bradyasystolic Cardiac Arrest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vancouver General Hospital (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Vancouver Coastal Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20F35869
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2003-09

CONDITIONS: Cardiac Arrest
Keywords: Heart Arrest; Cardiopulmonary Resuscitation; Aminophylline; Bradycardia; Humans; Emergency Medical Services
MeSH Terms: conditions — Heart Arrest; Bradycardia | interventions — Aminophylline

INTERVENTIONS:
Drug: Aminophylline (250mg IV +/- a second dose of 250mg IV)

SUMMARY:
The purpose of this study is to evaluate the effect of aminophylline in patients with out-of-hospital bradyasystolic cardiac arrest.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest treated by emergency medical services has an estimated incidence of 54.99 per 100,000 person years, which translates to some 155,000 episodes annually in the United States. Bradyasystole is the first recorded rhythm in up to 52 percent of cardiac arrests, and many additional patients with an initial cardiac arrest rhythm of ventricular fibrillation deteriorate to bradyasystole after defibrillation efforts. Survival to hospital discharge occurs in less than 3 percent of patients presenting with bradyasystole; however, due to its frequency, this rhythm accounts for over 17 percent of all cardiac arrest survivors. As a result, even a small improvement in survival from bradyasystolic cardiac arrest would result in thousands of lives saved annually.

Adenosine is an endogenous purine nucleoside that depresses the sinoatrial node, blocks atrioventricular conduction, inhibits the pacemaker activity of the His-Purkinje system and attenuates the effects of catecholamines. Since adenosine is produced and released by myocardial cells during ischemia and hypoxia, it may be a reversible factor in the etiology or perpetuation of bradyasystole. Aminophylline is a competitive antagonist of adenosine. The use of aminophylline for bradycardia and heart block has been described, and a number of anecdotal reports and small studies have been published on the use of aminophylline in cardiac arrest. We undertook this study to evaluate the effect of aminophylline during cardiopulmonary resuscitation (CPR) of patients with out-of-hospital bradyasystolic cardiac arrest unresponsive to initial therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest
* Bradyasystole either as the presenting rhythm or as a rhythm developing during the course of the resuscitation
* Endotracheally intubated and ventilated with 100% oxygen
* Intravenous (IV) access established
* Bradyasystolic without palpable pulses after 1 mg of epinephrine and 3 mg of atropine.

Exclusion Criteria:

* A do-not-resuscitate directive
* Pregnancy
* Evidence of hemorrhage, trauma or hypothermia as a cause of the cardiac arrest
* Renal dialysis
* Theophylline hypersensitivity
* Patients taking an oral theophylline product
* Resuscitations directed by a paramedic student under practicum supervision

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 966
Dates: Start 2001-01; Study Completion 2004-07

PRIMARY OUTCOMES:
The return of spontaneous circulation (ROSC), defined as the development of a palpable pulse of any duration.

SECONDARY OUTCOMES:
Maximum duration of ROSC (the duration of the longest episode of sustained pulse return)
ROSC duration by survival analysis
Survival to hospital admission
Survival to hospital discharge
Length of hospital stay
Non-sinus tachyarrhythmias in the first 24 hours after study drug administration
Seizures in the first 24 hours after study drug administration
Neurologic outcome
Proportion of subjects receiving one versus two doses of study drug
Proportion of subjects achieving ROSC with initial-rhythm bradyasystole versus bradyasystole which developed after paramedic arrival.

CONTACTS AND LOCATIONS:
Overall Officials: Riyad B Abu Laban, MD, MHSc, Principal Investigator — Department of Emergency Medicine, Vancouver General Hospital
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Abu-Laban RB, McIntyre CM, Christenson JM, van Beek CA, Innes GD, O'Brien RK, Wanger KP, McKnight RD, Gin KG, Zed PJ, Watts J, Puskaric J, MacPhail IA, Berringer RG, Milner RA. Aminophylline in bradyasystolic cardiac arrest: a randomised placebo-controlled trial. Lancet. 2006 May 13;367(9522):1577-84. doi: 10.1016/S0140-6736(06)68694-7. PMID 16698410